CLINICAL TRIAL: NCT07006883
Title: Effects of a Yoga Program on the Functionality of Individuals With Knee Osteoarthritis
Brief Title: Effects of a Yoga Program on the Functionality of Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Professor Phd, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 85065624.0.0000.5511
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercise group (Active Comparator): The program consists of warm-up, strengthening, and mobility exercises, based on functional movements that are typically challenging for individuals with knee osteoarthritis (KOA), in addition to balance exercises previously defined in a prior clinical trial.
  The program will be delivered in three phases:
  Phase 1 (weeks 0-2), Phase 2 (weeks 2-4), and Phase 3 (weeks 4-8).
  Every two weeks, participants will be reassessed to allow for potential adjustments aimed at promoting the progressive progression of the exercises.
  Interventions: Other: Therapeutic exercise
- Yoga therapeutic exercise (Experimental): The program was developed based on previous studies and considering the functional demands of each established position, as detailed in Tables 4, 5, and 6. The intervention will be structured into three phases:
  Phase 1 (weeks 0-2), Phase 2 (weeks 2-4), and Phase 3 (weeks 4-8). Every two weeks, participants will be reassessed to allow for potential adjustments, aiming to ensure the progressive progression of the exercises.
  Interventions: Other: Yoga therapeutic exercise

INTERVENTIONS:
Other: Therapeutic exercise — Therapeutic exercise focused on muscle strengthening, balance, and functional performance.
  Arms: Therapeutic exercise group
Other: Yoga therapeutic exercise — Yoga is a mind-body practice that integrates physical postures, breathing techniques, and mindfulness with the aim of improving physical function, balance, strength, mobility, and psychological well-being. I
  Arms: Yoga therapeutic exercise

SUMMARY:
There is a notable and emerging use of structured exercise programs incorporating Yoga for chronic musculoskeletal pain. However, regarding knee osteoarthritis (KOA), the effectiveness of Yoga remains uncertain to justify its inclusion in therapeutic exercise programs in routine clinical practice. Therefore, the aim of this project is to evaluate the effects of Yoga on functionality in individuals with KOA.

For this purpose, participants with KOA, including individuals of both sexes, aged 45 years or older, with a clinical diagnosis of KOA, will be randomly allocated using a random sequence generated by software, organized in six blocks of 24 codes, with an allocation ratio of 1:1, numbered sequentially from 1 to 126. Allocation will be concealed and performed after pre-intervention assessment and confirmation of eligibility criteria. Participants will be distributed into two groups: (1) Experimental group - Yoga (n = 45) and (2) Control group - therapeutic exercise (n = 45).

The intervention will last 8 weeks, with assessments conducted at baseline, after 4 weeks, and after 8 weeks of the intervention programs. The following outcome measures will be used: Knee Injury and Osteoarthritis Outcome Score (KOOS), Berg Balance Scale (BBS), Numeric Pain Rating Scale (NPRS), Pain Self-Efficacy Questionnaire (PSEQ), Global Perceived Effect Scale (GPE), 30-Second Sit-to-Stand Test (30s-STS), Timed Up and Go Test (TUG), and Maximal Voluntary Isometric Contraction (MVIC).

Data analysis will include a normality test to verify the distribution of the data, followed by the appropriate statistical tests for intra- and intergroup comparisons. The comparisons will consider two factors: time and group. A significance level of 5% (p < 0.05) will be adopted for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of knee osteoarthritis (knee pain for > 3 months)
* Morning stiffness <30 minutes
* Crepitus
* Bone tenderness, and absence of palpable heat and/or diagnosis established radiographically (determined by Kellgren and Lawrence grade 1 to 3 on a scale 1 up to 4)

Exclusion Criteria:

* Bilateral hip or KOA
* Severe osteoporosis
* Fibromyalgia
* Clinical history of tumors or cancer
* Active inflammatory joint diseases (rheumatoid arthritis, gout), undergoing any joint replacement of the lower extremity
* Neurological diseases (Parkinson's disease, Stroke, Multiple Sclerosis, muscular dystrophies, neuromotor disease, Alzheimer's disease)
* Infected wounds or osteomyelitis in the knee region
* Deep vein thrombosis or thrombophlebitis, sensory changes in the lower limbs
* A cognitive and cardiopulmonary impairment that may prevent or limit the performance of exercises
* Use of a walking assistance device, history of recent trauma to the knee
* Be performing or having prior any form of treatment involving physiotherapy, intra-articular corticosteroids, anti-inflammatories, opioid medication, or chondroprotective in the six months before the start of interventions

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-01-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Functional disability | Change from Baseline, after 4 weeks of intervention and 8 weeks after the end of the intervention.
  Knee Injury and Osteoarthritis Outcome Score (KOOS). It aims to evaluate the domains of pain, symptoms, activities of daily living, function related to recreation and sports, and quality of life related to the knee. Totaling 42 items, each item must be answered using a Likert scale that ranges from 0 (best score) to 4 (worst score), and the score for each subscale ranges from 0 (worst score) to 100 (best score).

SECONDARY OUTCOMES:
Numerical Pain Scale | Change from Baseline, after 4 weeks of intervention and 8 weeks after the end of the intervention.
  The Numerical rating pain scale, a simple, easily administered scale evaluates the perceived intensity of pain, using an 11-point scale from 0, representing 'no pain', to 10, which is the 'worst possible pain'.
Functional self-perception | Change from Baseline, after 4 weeks of intervention and 8 weeks after the end of the intervention.
  Pain self-efficacy questionnaire, structured into 10 items where each item is evaluated by selecting a number on a 7-point numerical scale (scores from 0 to 6), where 0 means "not at all confident" and 6 means "completely confident". The items cover different functions, from work, social activities, domestic tasks and coping with pain without medication. A total score is calculated from the sum of the scores for each of the 10 items, producing a total score that ranges from 0 to 60. Higher scores reflect stronger self-efficacy beliefs.
Global Perception of Change scale | Change from Baseline, after 4 weeks of intervention and 8 weeks after the end of the intervention.
  The perception of the global effect of the treatment by the research participant will be evaluated by the Global Perception of Change scale. The Global Perception of Change scale is a direct scale on the patient's self-perception when the intervention is performed. This scale consists of 11 points, ranging from -5 (worsening compared to the start of treatment), 0 (neutral) and +5 (improvement compared to the start of treatment), using the Portuguese version.
Dynamic balance | Change from Baseline, after 4 weeks of intervention and 8 weeks after the end of the intervention.
  Iimed up and go test, research participants will be instructed to get up from a chair, walk 3 meters comfortably and safely, come back and sit down in the chair. The time taken to complete this task will be measured using a stopwatch that will be started after the verbal command 'go' and stopped when the participant returns to the initial sitting position. A first attempt will be made to familiarize the participant with the procedure. Two assessments will then be carried out. The average of the two assessments will be recorded for later data analysis.
Maximum voluntary isometric contraction | Change from Baseline, after 4 weeks of intervention and 8 weeks after the end of the intervention.
  manual dynamometer portable (Lafayette Manual Muscle System, Modelo 01165, Lafayette Instrument Company, Lafayette, IN). Four 5-second readings will be taken during maximal voluntary isometric contraction (MVIC) with a 30-second rest period between contractions. The first CIVM will familiarize the volunteer with carrying out the task. A new set of readings will be taken if a volunteer can perform three contractions with at least 10% variability. Strong and constant verbal stimuli will be used throughout the test. Always with the research participants' hands positioned crossed on the chest. Thus, bilateral assessments of the muscles, quadriceps, and gluteus medius will be carried out. The order of CIVM readings will be randomized to avoid collection bias. The research participant will remain in lateral decubitus with a pillow positioned between the legs, with the limb to be tested superiorly in a neutral position.
Stand Test | Change from Baseline, after 4 weeks of intervention and 8 weeks after the end of the intervention.
  The 30-Second Chair Stand Test (30s-CST) assesses physical function and is recommended by OARSI for individuals with knee osteoarthritis (KOA). The participant performs as many sit-to-stand repetitions as possible in 30 seconds, using a 43 cm-high, straight-backed chair without armrests, placed against a wall. The starting position is seated, feet flat, hip-width apart, and arms crossed over the chest. Two to three practice repetitions are recommended. If unable to stand independently, participants may use hand support or a mobility aid, with score adjustments. The same chair must be used for all assessments.
functional balance | Change from Baseline, after 4 weeks of intervention and 8 weeks after the end of the intervention.
  The Berg Balance Scale (BBS) is a functional assessment of static and dynamic balance. It consists of 14 items, each scored on a 4-point Likert scale, with a total score ranging from 0 to 56 points. Risk of falls is classified as follows:
  0 to 20: high risk of falls, 21 to 40: moderate risk of falls, and 41 to 56: low risk of falls. The Brazilian Portuguese version of the BBS has been translated, cross-culturally adapted, and validated, demonstrating adequate levels of reliability and measurement consistency.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No